CLINICAL TRIAL: NCT07330128
Title: Parent/Caregiver-Involved Nutrition Education in Down Syndrome: A Single-Group Pre-Post Quasi-Experimental Study
Brief Title: Caregiver-Involved Nutrition Education in Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hülya YILMAZ ÖNAL (Other)
Responsible Party: Sponsor-Investigator, Hülya YILMAZ ÖNAL, Associate Professor, Istanbul Medeniyet University
Organization: Istanbul Medeniyet University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2024/1, dated 23 January 2024
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Down Syndrome
Keywords: Health Education; Nutritional Status; Anthropometry
MeSH Terms: conditions — Down Syndrome; Health Education

STUDY DESIGN:
Intervention Model Description: Single-arm pre-post design (one group assessed before and after an 8-week online nutrition education program)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutrition Education (Caregiver-Involved) (Experimental): Participants received an 8-week online nutrition education program. Individuals with Down syndrome attended weekly sessions (~15 minutes) focusing on understanding food groups, adopting healthy eating principles, reducing sugary/packaged foods, increasing daily physical activity, and emphasizing adequate daily water intake. Caregivers received four modules (~30 minutes each) covering healthy eating principles, food groups, physical activity, common comorbidities and metabolic changes in Down syndrome, and key considerations in nutrition therapy. Sessions were delivered via live video conferencing with slide-based materials shared during sessions and sent afterward via online messaging.
  Interventions: Behavioral: Caregiver-Involved Nutrition Education

INTERVENTIONS:
Behavioral: Caregiver-Involved Nutrition Education — An 8-week online nutrition education program delivered via live video conferencing with slide-based materials shared during sessions and sent afterward to caregivers.

SUMMARY:
This single-arm, quasi-experimental pre-post study evaluated an 8-week online nutrition education program for individuals with Down syndrome and their caregivers in Ataşehir, Istanbul, Türkiye. Thirty-one individuals with Down syndrome and 31 caregivers (n=62) completed the program. Dietary behaviors, 3-day dietary intake, anthropometric measurements, and caregiver nutrition literacy were assessed before and after the intervention.

DETAILED DESCRIPTION:
Participants were recruited through the Turkey Down Syndrome Association (Ataşehir, Istanbul). Eligible participants were individuals with Down syndrome who could express preferences and caregivers with sufficient digital skills to complete online procedures. Although 39 individuals initially agreed to participate, the study was completed with 31 individuals with Down syndrome and their caregivers (n=62) after exclusions for eligibility and continuity.

Data were collected using a Down Syndrome Individual Information Form, the Nutrition Behavior Scale, a 3-day dietary intake record (including one weekend day; analyzed in BeBİS), a Caregiver Information Form, the Adult Nutrition Literacy Assessment Tool, and Down syndrome-specific growth charts (Zemel et al., 2015; 2-20 years).

The intervention consisted of an 8-week basic nutrition education program delivered via live video conferencing. Individuals with Down syndrome received weekly sessions of approximately 15 minutes focusing on food groups, healthy eating principles, reducing sugary/packaged foods, increasing daily physical activity, and adequate water intake. Caregivers received four modules of approximately 30 minutes covering healthy eating principles, food groups, physical activity, common comorbidities and metabolic changes in Down syndrome, and key considerations in nutrition therapy. Illustrated and graphical slide materials were shared during sessions and sent to caregivers afterward via online messaging.

ELIGIBILITY:
Inclusion Criteria:

Volunteered to participate and provided informed consent (caregiver/parent consent).

Individuals with Down syndrome who were able to express their preferences. Caregivers/parents with sufficient digital knowledge and skills to participate in online procedures and training sessions.

Exclusion Criteria:

* Individuals with Down syndrome and/or caregivers/parents who did not have sufficient digital knowledge and skills to participate in online procedures.

Individuals with Down syndrome and/or caregivers/parents who did not maintain continuity in the study (e.g., did not complete the intervention and/or pre-/post-assessments).

Ages: 6 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-02-27 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Dietary behavior (Nutrition Behavior Scale score) | Baseline (pre-intervention) and immediately after the 8-week education program.
  Change in dietary behavior score measured using the Nutrition Behavior Scale (total score range -14 to +14; converted to a 0-100% healthy consumption score).

SECONDARY OUTCOMES:
Dietary intake from 3-day diet records (energy and selected nutrients) | Baseline (pre-intervention) and immediately after the 8-week education program.
  Change in daily energy and nutrient intakes derived from 3-day dietary intake records (including one weekend day) and analyzed using the BeBİS nutrition analysis software (e.g., energy, protein, dietary fiber, selected vitamins/minerals, n-3 and n-6 fatty acids).
BMI | Baseline (pre-intervention) and immediately after the 8-week education program.
  Change in body weight and BMI
Anthropometric measurements | Baseline (pre-intervention) and immediately after the 8-week education program.
  Change in anthropometric measurements (e.g., age-appropriate interpretation using Down syndrome-specific growth charts where applicable).

CONTACTS AND LOCATIONS:
Overall Officials: Hülya Yılmaz Önal, Assoc. Prof., Principal Investigator — stanbul Medeniyet University, Department of Nutrition and Dietetics
Locations (1):
- Turkey Down Syndrome Association (, Istanbul, Turkey (Türkiye)